CLINICAL TRIAL: NCT06352086
Title: Understanding Visual Processing After Occipital Stroke
Status: Withdrawn | Type: Observational
Why Stopped: Study was never officially approved by IRB and never open to enrollment. Submission withdrawn due to lack of funding.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Krystel Huxlin, James V. Aquavella Professor of Ophthalmology, Associate Chair for Research, Dept. Ophthalmology, University of Rochester
Other Study IDs: STUDY00009227
Record Dates: First submitted 2024-04-01; First posted 2024-04-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Vision Loss Partial; Vision; Loss, Both Eyes; Hemianopia, Homonymous; Hemianopia; Quadrantanopia; Stroke, Ischemic; Stroke - Occipital Infarction; Cortical Blindness; Occipital Lobe Infarct; Peripheral Visual Field Defect of Both Eyes
Keywords: Occipital stroke; Vision loss after stroke; Vision recovery; Vision restoration; Partial vision loss; vision loss
MeSH Terms: conditions — Blindness; Hemianopsia; Ischemic Stroke; Blindness, Cortical; Vision Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to investigate how visual orientation discrimination and metacognition (i.e., perceptual confidence) are affected by occipital stroke that causes hemianopia and quadrantanopia in adults. This research will provide insight as to how the residual visual system, which not directly damaged by the occipital stroke, processes orientation (assayed in terms of orientation discrimination) and metacognition (by measuring perceptual confidence for orientation discrimination). These measures will be used to refine computational models that attempt to explain how the brain copes with loss of primary visual cortex (V1) as a result of stroke. This knowledge is essential to devise more effective visual rehabilitation therapies for patients suffering from occipital strokes.

ELIGIBILITY:
Inclusion Criteria:

* Residents of the United States or Canada
* MRI and/or CT scans showing unilateral stroke or stroke-like damage to primary visual cortex or its immediate afferent white matter sustained 1-year or more prior to enrollment
* Reliable visual field defects in both eyes as measured by Humphrey, Macular Integrity Assessment (MAIA), Goldmann, and/or equivalent perimetry. This deficit must be large enough to enclose a 5-deg diameter visual stimulus.
* Ability to fixate on visual targets reliably for 1000ms (as demonstrated by visual fields, and verified in study participation)
* Willing, able, and competent to provide informed consent
* Cognitively able to understand and respond to written and oral instructions in English

Exclusion Criteria:

* Past or present ocular disease interfering with visual acuity
* Corrected vision worse than 20/40 in either eye
* Presence of damage to the dorsal Lateral Geniculate Nucleus
* Diffuse, whole brain degenerative processes
* Brain damage deemed by study staff to potentially interfere with testing ability or outcome measures
* Documented history of traumatic brain injury
* Documented history of drug/alcohol abuse
* Current use neuroactive
* Cognitive or seizure disorders
* Subjects with one-sided attentional neglect

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will all be individuals who have sustained partial vision loss after an occipital lobe stroke.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Orientation discrimination threshold | Baseline
  Assessment of Static Orientation Discrimination.
  For each subject, the investigators will measure the ability to correctly identify the orientation of non-moving visual stimuli that vary in degree of angle tilt to the right or left of vertical. The investigators will measure the degree of angle tilt that can be reliably detected at a 72-75% correct level of performance. Tilt difference from vertical will vary between 80° (maximum) and 0.1° (minimum) based on subject performance and an adaptive staircase that will change tilt magnitude depending on subject performance, increasing the tilt (making the task easier) for each incorrect answers and decreasing tilt (making the task harder) after a number of correct answers in a row.
Perceptual Confidence in Orientation Discrimination | Baseline
  Assessment of Metacognition (i.e., perceptual confidence) in Orientation Discrimination.
  For each subject, the investigators will measure their confidence in identifying an object's tilt to the right or left of vertical. A running tally of 'response points' will be collected during the orientation testing. Points will be awarded for each response on a scale, with the highest points awarded for "correct discrimination & high confidence", intermediate points awarded for "correct discrimination & low confidence", followed by "incorrect discrimination & low confidence" and with points subtracted for "incorrect discrimination & high confidence". Total points will be recorded for each test, with the patient asked to accumulate the highest number of points they can during the task.